CLINICAL TRIAL: NCT02199041
Title: Combined T Cell Depleted Haploidentical Peripheral Blood Stem Cell and Unrelated Umbilical Cord Blood Transplantation in Patients With Hematologic Malignancies Using a Total Lymphoid Irradiation Based Preparative Regimen
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was halted early due to slow accrual.
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAPCORD; NCI-2014-00526 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2014-07-09; First posted 2014-07-24 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2017-08

CONDITIONS: Hematological Malignancies
Keywords: Cord Blood; Haploidentical; Reduced Intensity Regimen
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Cyclophosphamide; Thiotepa; fludarabine; fludarabine phosphate; Melphalan; Mesna; Granulocyte Colony-Stimulating Factor; Filgrastim; Mycophenolic Acid; Tacrolimus; Methylprednisolone; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment (Experimental): Interventions: cyclophosphamide, thiotepa, fludarabine, melphalan, mesna, granulocyte colony-stimulating factor (G-CSF), mycophenolate mofetil, tacrolimus, methylprednisolone, total lymphoid irradiation, and lymphocyte infusions.
  Cells for infusion are prepared using the CliniMACS System.
  Interventions: Drug: Cyclophosphamide; Drug: Thiotepa; Drug: Fludarabine; Drug: Melphalan; Drug: Mesna; Biological: G-CSF; Drug: Mycophenolate mofetil; Drug: Tacrolimus; Drug: Methylprednisolone; Radiation: Total lymphoid irradiation; Biological: Lymphocyte infusions; Device: CliniMACS

INTERVENTIONS:
Drug: Cyclophosphamide — Given by intravenous infusion as part of the preparative regimen.
  Other Names: Cytoxan
Drug: Thiotepa — Given by intravenous infusion as part of the preparative regimen.
  Other Names: Thioplex(R); TESPA; TSPA
Drug: Fludarabine — Given by intravenous infusion as part of the preparative regimen.
  Other Names: Fludara
Drug: Melphalan — Given by intravenous infusion as part of the preparative regimen.
  Other Names: L-phenylalanine mustard; Phenylalanine mustard; L-PAM; L-sarcolysin; Alkeran
Drug: Mesna — Mesna is generally dosed at approximately 25% of the cyclophosphamide dose. It is generally given intravenously prior to and again at 3, 6 and 9 hours following each dose of cyclophosphamide.
  Other Names: Mesnex
Biological: G-CSF — Given either by intravenous infusion or subcutaneously daily until absolute neutrophil count (ANC) >2000 for 3 consecutive days.
  Other Names: Granulocyte colony-stimulating factor (C-CSF); Filgrastim; Neupogen(R)
Drug: Mycophenolate mofetil — Given either orally or by intravenous infusion as part of the post-transplantation immunosuppression.
  Other Names: MMF; CellCept(R)
Drug: Tacrolimus — Given either orally or by intravenous infusion as part of the post-transplantation immunosuppression.
  Other Names: FK506; Prograf(R); Protopic(R)
Drug: Methylprednisolone — Given either intravenously or orally, if needed to treat graft-versus-host-disease (GVHD).
  Other Names: Medrol(R); Solu-Medrol
Radiation: Total lymphoid irradiation — TLI will be administered in divided fractions given at a minimum of 6 hours apart.
  Other Names: TLI
Biological: Lymphocyte infusions — Donors will undergo haploidentical mobilization with G-CSF. Cells will be collected by leukapheresis over two days, then processed using the investigational CliniMACS device and CD34 Microbead reagent as directed by the manufacturer.
  Other Names: Donor lymphocyte infusions; DLI
Device: CliniMACS — The mechanism of action of the CliniMACS Cell Selection System is based on magnetic-activated cell sorting (MACS). The CliniMACS device is a powerful tool for the isolation of many cell types from heterogeneous cell mixtures, (e.g. apheresis products). These can then be separated in a magnetic field using an immunomagnetic label specific for the cell type of interest, such as CD3+ human T cells.
  Other Names: Cell Selection System

SUMMARY:
In this study, participants with high-risk hematologic malignancies undergoing hematopoietic cell transplantation (HCT), who do not have a suitable human leukocyte antigen (HLA)-matched related/sibling donor (MSD), matched unrelated donor (MURD) or killer-immunoglobulin receptors (KIR) ligand mismatched haploidentical donor identified, will receive a combined T cell depleted (TCD) haploidentical peripheral blood stem cell (PBSC) and unrelated umbilical cord blood transplantation (UCBT) using a total lymphoid irradiation (TLI) based preparative regimen.

Primary objective:

* To estimate the incidence of donor derived neutrophil engraftment by day +42 post-transplant for participants with high-risk hematologic malignancies undergoing a total lymphoid irradiation (TLI)-based hematopoietic cell transplantation (HCT) using a T cell depleted (TCI) haploidentical donor peripheral blood stem cell (PBSC) donor combined with an unrelated umbilical cord blood (UCB) donor.

Secondary objectives:

* Estimate the incidence of malignant relapse, event-free survival (EFS), and overall survival (OS) at one-year post-transplantation.
* Estimate the incidence and severity of acute and chronic graft versus host disease (GVHD) in the first 100 days after transplantation.
* Estimate the incidence of secondary graft failure transplant related mortality (TRM) and transplant related morbidity in the first 100 days after HCT.

DETAILED DESCRIPTION:
Prior to stem cell infusion, participants will receive a preparative regimen of total lymphoid irradiation (TLI), fludarabine, cyclophosphamide, melphalan, and thiotepa to prepare their bone marrow. Thereafter, they will receive a hematopoietic cell graft from a haploidentical donor and an unrelated umbilical cord blood donor. Post-transplantation immunosuppressive treatment will include tacrolimus and mycophenolate mofetil.

ELIGIBILITY:
Inclusion Criteria-Transplant Recipient:

* Age less than or equal to 21 years old.
* Does not have a suitable matched related/sibling donor (MSD) or volunteer matched unrelated donor (MUD) available in the necessary time for stem cell donation.
* Has a suitable partially human leukocyte antigen (HLA)-matched (≥ 3 of 6) family member donor.
* Has a partially HLA-matched single umbilical cord blood (UCB) unit (≥ 4 of 6) with adequate cell dose. UCB units must fulfill eligibility as outlined in 21 CFR 1271 and agency guidance.
* High-risk hematologic malignancy.

  * High risk acute lymphocytic leukemia (ALL) in complete remission-1 (CR)1. [Examples include, but not limited to t(9;22), hypodiploid,, M2 or greater marrow at the end of induction, infants with mixed lineage leukemia (MLL) fusion or t(4;11)].
  * ALL in High risk CR2. [Examples include but not limited to t(9;22), bone marrow (BM) relapse <36 mo CR1, T-ALL, very early (< 6mo CR1) isolated central nervous system (CNS) relapse.]
  * ALL in CR3 or subsequent.
  * Acute myeloid leukemia (AML) in high risk CR1. [Examples include but not limited to preceding MDS, 5q-, -5, -7, FAB M6, FAB M7 not t(1;22), minimal residual disease (MRD) ≥ 5% on day 22 (AML08), M3 marrow after induction 1, M2 marrow after two cycles of induction, FLT3-ITD.]
  * AML in CR2 or subsequent.
  * Therapy related AML, with prior malignancy in CR > 12mo
  * Myelodysplastic syndrome (MDS), primary or secondary
  * Natural killer (NK) cell, biphenotypic, or undifferentiated leukemia in CR1 or subsequent.
  * Chronic myeloid leukemia (CML) in accelerated phase, or in chronic phase with persistent molecular positivity or intolerance to tyrosine kinase inhibitor.
  * Hodgkin lymphoma in CR2 or subsequent after failure of prior autologous hematopoietic cell transplantation (HCT), or unable to mobilize stem cells for autologous HCT.
  * Non-Hodgkin lymphoma in CR2 or subsequent.
  * Juvenile myelomonocytic leukemia (JMML).
  * Refractory hematologic malignancies [ALL, AML, chronic myeloid leukemia (CML) in blast crisis, Hodgkin or non-Hodgkin lymphoma] due to chemoresistant relapse or primary induction failure.
  * All patients with evidence of CNS leukemia must be treated and be in CNS CR to be eligible for study.
* Patient must fulfill pre-transplant evaluation:

  * Cardiac Function: Left ventricular ejection fraction (LVEF) ≥ 40% or shortening fraction (SF) ≥ 25%.
  * Creatinine clearance (CrCL) or glomerular filtration rate (GFR) ≥ 50 ml/min/1.73m2.
  * Forced vital capacity (FVC) ≥ 50% of predicted value or pulse oximetry (Pox) ≥ 92% on room air.
  * Karnofsky or Lansky performance score ≥ 50.
  * Bilirubin ≤ 3 times the upper limit of normal for age.
  * Alanine aminotransferase (ALT) ≤ 5x the upper limit of normal for age.
  * Aspartate aminotransferase (AST) ≤ 5x the upper limit of normal for age.

Exclusion Criteria - Transplant Recipient:

* Patient has a suitable MSD, volunteer matched unrelated donor (MURD), or killer-immunoglobulin receptors (KIR) mismatched haploidentical donor available in the necessary time for stem cell donation.
* Patient has any other active malignancy other than the one for which HCT is indicated.
* Patient is pregnant as confirmed by positive serum or urine pregnancy test within 14 days prior to enrollment.
* Patient is breast feeding.
* Patient has Down Syndrome.
* Patient has a current uncontrolled bacterial, fungal, or viral infection per the judgment of the principal investigator.

Inclusion criteria - haploidentical donor

* At least single haplotype matched (≥ 3 of 6) family member
* At least 18 years of age.
* Human immunodeficiency virus (HIV) negative.
* Not pregnant as confirmed by negative serum or urine pregnancy test within 14 days prior to enrollment (if female).
* Not breast feeding.
* Regarding eligibility, is identified as either:

  * Completed the process of donor eligibility determination as outlined in 21 CFR 1271 and agency guidance; OR
  * Does not meet 21 CFR 1271 eligibility requirements, but has a declaration of urgent medical need completed by the principal investigator or physician sub-investigator per 21 CFR 1271.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2014-07-11 (Actual); Primary Completion 2017-05-23 (Actual); Study Completion 2017-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Triplett, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twelve participants meeting eligibility criteria and 12 of their blood donors were enrolled at St. Jude Children's Research Hospital between July 2014 and January 2015.
Pre-assignment Details: The 12 enrolled blood donors did not undergo transplantation and are therefore not included in the results reported here.
Groups:
- Treatment: Interventions: cyclophosphamide, thiotepa, fludarabine, melphalan, mesna, granulocyte colony-stimulating factor (G-CSF), mycophenolate mofetil, tacrolimus, methylprednisolone, total lymphoid irradiation, and lymphocyte infusions.
  Cells for infusion are prepared using the CliniMACS System.
  Prior to stem cell infusion, participants receive a preparative regimen of total lymphoid irradiation (TLI), fludarabine, cyclophosphamide, melphalan, and thiotepa to prepare their bone marrow. Thereafter, they will receive a hematopoietic cell graft from a haploidentical donor and an unrelated umbilical cord blood donor. Post-transplantation immunosuppressive treatment will include tacrolimus and mycophenolate mofetil.
Period: Overall Study
Arm/Group | Treatment
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment: Interventions: cyclophosphamide, thiotepa, fludarabine, melphalan, mesna, G-CSF, mycophenolate mofetil, tacrolimus, methylprednisolone, total lymphoid irradiation, and lymphocyte infusions.
  Cells for infusion are prepared using the CliniMACS System.
  Prior to stem cell infusion, participants receive a preparative regimen of total lymphoid irradiation (TLI), fludarabine, cyclophosphamide, melphalan, and thiotepa to prepare their bone marrow. Thereafter, they will receive a hematopoietic cell graft from a haploidentical donor and an unrelated umbilical cord blood donor. Post-transplantation immunosuppressive treatment will include tacrolimus and mycophenolate mofetil.
Arm/Group | Treatment
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.7 (7.5)
Age, Continuous [Median (Full Range); unit: years] | 5.0 [0.7 to 20.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — NOS = Not Otherwise Specified
  Participants
    Ethnicity: NOS Spanish, Hispanic, Latino | 1
    Ethnicity: Non Spanish Speaking, Non Hispanic | 8
    Ethnicity: Puerto Rican | 1
    Ethnicity: South or Central American | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — NOS = Not Otherwise Specified
  Participants
    Race: Black | 3
    Race: Multiple Race (NOS) | 1
    Race: White | 8
Diagnosis [Count of Participants; unit: Participants] — AL = Acute Leukemia; BM = Bone Marrow
  Participants
    Acute Erythroleukemia, FAB M6, BM | 1
    AL, Lymphoblastic, Pre-B, BM | 2
    AL, Lymphoblastic, Pre-T Cell, BM | 1
    AL, Megakaryoblastic, FAB M7, BM | 2
    AL, Monocytic, FAB M5, BM | 1
    AL, Myeloid, Minimal Differentiation, FAB M0, BM | 1
    AL, Myeloid, NOS, BM | 2
    AL, Myeloid, With Maturation, FAB M2, BM | 1
    Lymphoma, Non-Hodgkin's, Anaplastic Large Cell | 1
Disease Status at HSCT [Count of Participants; unit: Participants] — Complete remission (CR) defined as less than 5 percent leukemia blasts in a bone marrow with evidence of hematopoietic recovery. Relapse is defined as return of 5 percent leukemia blasts or more in a bone marrow after previous achieving CR. Refractory is defined as never achieving CR despite therapy, also known as induction failure. The disease status worsens going down the list with CR1 indicating the best prognosis and Relapse 2 the worst prognosis.
  Participants
    CR1 | 2
    CR2 | 3
    CR3 | 2
    Refractory | 4
    Relapse 2 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Neutrophil Engraftment
Description: Neutrophil engraftment is defined as absolute neutrophil count (ANC) recovery of ≥ 0.5 x 10^9/L (500/mm^3) for three consecutive laboratory values obtained on different days (derived from either donor). Date of engraftment is the date of the first of the three consecutive laboratory values. The number of patients engrafted by day +42 post-transplant is provided.
Time Frame: Until day 42 post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
Participants | 11

2. Secondary Outcome: Number of Participants With Malignant Relapse
Description: Relapse was evaluated using standard World Health Organization (WHO) criteria for each disease. The estimate of cumulative incidence of relapse will be estimated using Kalbfleisch-Prentice method. Relapse defined as the recurrence of original disease. Death is the competing risk event. The analysis will be implemented using Statistical Analysis System (SAS) macro (bmacro252-Excel2007\cin).
  Due to the early close of the study, a small number of patients were enrolled. Subsequently, the number of patients who experienced malignant relapse is provided
Time Frame: One year after transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
Participants | 7

3. Secondary Outcome: Number of Participants With Event-free Survival (EFS)
Description: The Kaplan-Meier estimate of EFS with relapse, death due to any cause and graft failure as events along with their standard errors will be calculated using the SAS macro (bmacro251-Excel2007\kme) available in the Department of Biostatistics at St. Jude, where EFS = min (date of last follow-up, date of relapse, date of graft failure, date of death due to any cause) - date of transplant, and all participants surviving at the time of analysis without events will be censored. The number of participants who did not experience any of these events through one year post-transplant is given.
  Due to the early close of the study, a small number of patients were enrolled. Subsequently, the number of patients who did not experience any events defined above is provided.
Time Frame: One year after transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
Participants | 4

4. Secondary Outcome: Number of Participants With Overall Survival (OS)
Description: The Kaplan-Meier estimate of OS with relapse, death due to any cause and graft failure as events along with their standard errors will be calculated using the SAS macro (bmacro251-Excel2007\kme) available in the Department of Biostatistics at St. Jude, where OS = min (date of last follow-up, date of death) - date of hematopoietic cell transplantation (HCT) and all participants surviving after 1 year post-transplant will be considered as censored.
  Due to the early close of the study, a small number of patients were enrolled. Subsequently, the number of patients who did not die at 1 year post-transplant is provided.
Time Frame: One year after transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
Participants | 6

5. Secondary Outcome: Number of Participants by Severity With Acute Graft Versus Host Disease (GVHD) in the First 100 Days After HCT
Description: Cumulative incidence of acute GVHD was estimated using Kalbfleisch-Prentice method. Death is the competing risk event. SAS macro (bmacro252-Excel2007\cin) available at St. Jude was used for analysis. Severity of GVHD and stage were determined using the Clinical Oncology Group (COG) Stem Cell Committee Consensus Guidelines for establishing organ stage and overall grade of acute GVHD. Participants are graded on a scale from I to IV, with I being mild and IV being severe.
  Overall Clinical Grade (based on the highest stage obtained):
  Grade 0: No stage 1-4 of any organ. Grade I: Stage 1-2 skin and no liver or gut involvement. Grade II: Stage 3 skin, or Stage I liver involvement, or Stage 1 gastrointestinal (GI).
  Grade III: Stage 0-3 skin, with Stage 2-3 liver, or Stage 2-3 GI. Grade IV: Stage 4 skin, liver or GI involvement.
  Due to early close of study, a small number of patients were enrolled. The number of patients who experienced acute GVHD is provided.
Time Frame: 100 days after transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
Participants
  No Acute GVHD | 8
  Grade I | 0
  Grade II | 1
  Grade III | 2
  Grade IV | 1

6. Secondary Outcome: Number of Participants by Severity With Chronic Graft Versus Host Disease (GVHD) in the First 100 Days After HCT
Description: Cumulative incidence of acute and chronic GVHD was estimated using Kalbfleisch-Prentice method. Death is competing risk event. SAS macro (bmacro252-Excel2007\cin) available St. Jude was used for such analysis. Severity of chronic GVHD was evaluated using National Institutes of Health (NIH) Consensus Global Severity Scoring. Mild is considered a better outcome with severe being the worst.
  Criteria for grading chronic GVHD:
  Mild: 1-2 organs/sites, maximum organ score of 1, and lung score of 1. Moderate: 3 or more organs/sites and maximum organ score of 1 and lung score of 1, OR at least 1 organ/site and maximum organ score of 2 and lung score of 1. Severe: At least 1 organ/site and maximum organ score of 3 and lung score of 2-3.
  Due to the early close of the study, a small number of patients were enrolled. Subsequently, the number of patients who experienced chronic GVHD is provided.
Time Frame: 100 days after transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
Participants
  No Chronic GVHD | 11
  Mild | 0
  Moderate | 0
  Severe | 1

7. Secondary Outcome: Number of Participants With Secondary Graft Failure
Description: The cumulative incidence of secondary graft failure will be estimated using the Kalbfleisch-Prentice method. Deaths due to toxicity and relapse before day 100 are the competing events.
  Secondary graft failure or graft rejection will be defined as no evidence of donor chimerism by umbilical cord blood (UCB) and/or haploidentical donor (<10%), or too few cells to perform adequate chimerism analysis, in research participants with prior neutrophil engraftment.
  Due to the early close of the study, a small number of patients were enrolled. Subsequently, the number of patients who experienced secondary graft failure is provided.
Time Frame: 100 days after transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
Participants | 0

8. Secondary Outcome: Number of Participants With Transplant-related Mortality (TRM)
Description: TRM is any death in remission and related to protocol therapy. The cumulative incidence of TRM was estimated using the Kalbfleisch-Prentice method. Deaths before day 100 because of other reasons are the completing events.
  Due to the early close of the study, a small number of patients were enrolled. Subsequently, the number of patients who experienced TRM is provided.
Time Frame: 100 days after transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
Participants | 0

9. Secondary Outcome: Number of Participants With Transplant-related Morbidity
Description: Any patient who had adverse events listed either as probable or definite in the first 100 days post-transplant are counted as transplant-related morbidity. The cumulative incidence of transplant-related morbidity will be estimated using the Kalbfleisch-Prentice method. Deaths before day 100 are the competing risk events.
  Due to the early close of the study, a small number of patients were enrolled. Subsequently, the number of patients who experienced at least one-transplant-related morbidity is provided.
Time Frame: 100 days after transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
Participants | 12

ADVERSE EVENTS:
Time Frame: Adverse events were collected from participants beginning with the on-study date through one year post-transplantation.
Description: Adverse events were monitored for donors beginning with the on-study date through one year post-transplantation.
Groups:
- Blood Donors: Blood donors were enrolled on the study to provide cells for transplantation used in the Treatment Arm.
Arm/Group | Treatment | Blood Donors
All-Cause Mortality (participants affected / at risk) | 6/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 5/12 | 0/12
Other Adverse Events (participants affected / at risk) | 12/12 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=12) | Blood Donors (N=12)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 1 (1) | 0 (0)
Thrombotic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Fever without Neutropenia (General disorders) | 1 (1) | 0 (0)
Weight Loss (Investigations) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Infection, Enterobacter Cloacae, Blood (Infections and infestations) | 1 (1) | 0 (0)
Infection, Fungal and Viral, Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Infection, Staphylococcus Aureus, Blood (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia, Staph Aureus (Infections and infestations) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=12) | Blood Donors (N=12)
Acute Infusion Reaction, Stem Cells (Immune system disorders) | 2 (2) | 0 (0)
Allergic Reaction, Platelet Transfusion (Immune system disorders) | 1 (1) | 0 (0)
Allergy to Diary Product (Disorder) (Immune system disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 6 (8) | 0 (0)
Left Ventricular Cardiac Dysfunction (Disorder) (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 3 (4) | 0 (0)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Weight Loss (Investigations) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash, Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Colitis (Disorder) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypernatremic Dehydration (Disorder) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Disorder) (Gastrointestinal disorders) | 2 (2) | 0 (0)
Veno-Occlusive Disease, Hepatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cellulitis, Gastrostomy Site (Infections and infestations) | 1 (1) | 0 (0)
Fever without Neutropenia (Infections and infestations) | 1 (1) | 0 (0)
Febrile Neutropenia (Infections and infestations) | 12 (13) | 0 (0)
Hepatitis (Infections and infestations) | 1 (1) | 0 (0)
Infection, Adenovirus, Respiratory Tract (Infections and infestations) | 1 (1) | 0 (0)
Infection, Adenovirus, Stool (Infections and infestations) | 4 (5) | 0 (0)
Infection, BK Virus, Blood (Infections and infestations) | 1 (1) | 0 (0)
Infection, BK Virus, Urine (Infections and infestations) | 1 (1) | 0 (0)
Infection, CMV, Respiratory/Nasopharynx (Infections and infestations) | 1 (1) | 0 (0)
Infection, Candida Albicans, Oral Mucosa (Infections and infestations) | 1 (1) | 0 (0)
Infection, Candida Lipolytica, Oral Mucosa (Infections and infestations) | 1 (1) | 0 (0)
Infection, Clostridium Difficile Colitis (Infections and infestations) | 1 (1) | 0 (0)
Infection, Clostridium Difficile, Stool (Infections and infestations) | 1 (1) | 0 (0)
Infection, Cytomegalovirus, Blood (Infections and infestations) | 1 (1) | 0 (0)
Infection, Due to Klebsiella, Bone Marrow Site (Infections and infestations) | 1 (1) | 0 (0)
Infection, Enterobacter Asburiae, Blood (Infections and infestations) | 1 (1) | 0 (0)
Infection, Enterobacter Cloacae, Blood (Infections and infestations) | 1 (2) | 0 (0)
Infection, Enterobacter asburiae and Coagulase Negative Staphylococcus, Gastrostomy Wound Site (Infections and infestations) | 1 (1) | 0 (0)
Infection, Fungal, Liver (Infections and infestations) | 1 (1) | 0 (0)
Infection, Herpes Simplex Virus, Oral Mucosa (Infections and infestations) | 1 (1) | 0 (0)
Infection, Human Herpes Simplex Virus, Oral (Infections and infestations) | 1 (1) | 0 (0)
Infection, Human Herpes Virus 6, Blood (Infections and infestations) | 8 (8) | 0 (0)
Infection, Human Herpes Virus 6, Cerebrospinal Fluid (Infections and infestations) | 1 (1) | 0 (0)
Infection, Klebsiella pneumoniae, Colon (Infections and infestations) | 1 (1) | 0 (0)
Infection, Malassezia Furfur, Blood (Infections and infestations) | 1 (1) | 0 (0)
Infection, Norovirus, Stool (Infections and infestations) | 1 (1) | 0 (0)
Infection, Pediococcus Pentosaceua (Infections and infestations) | 1 (1) | 0 (0)
Infection, Presumed Viral, Oral Mucosa (Infections and infestations) | 1 (1) | 0 (0)
Infection, Rotavirus, Stool (Infections and infestations) | 3 (6) | 0 (0)
Infection, Staphylococcus Epidermidis, Blood (Infections and infestations) | 1 (1) | 0 (0)
Reactivation, Human Herpes Virus 6, Blood (Infections and infestations) | 1 (1) | 0 (0)
Hypoxia (Infections and infestations) | 1 (1) | 0 (0)
Ulceration, Larynx (Infections and infestations) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Insufficiency (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal, Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Engraftment Syndrome (Immune system disorders) | 2 (2) | 0 (0)
Pain, Abdomen (General disorders) | 2 (2) | 0 (0)
Pain, Neuropathic, Legs and Feet, Bilateral (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was halted early due to slow accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan: v. 0.0 - Initial (2014-02-26): https://cdn.clinicaltrials.gov/large-docs/41/NCT02199041/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: v. 0.1 (2014-10-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT02199041/Prot_SAP_001.pdf
  • Study Protocol and Statistical Analysis Plan: v. 1.0 (2016-05-04): https://cdn.clinicaltrials.gov/large-docs/41/NCT02199041/Prot_SAP_002.pdf
  • Study Protocol and Statistical Analysis Plan: v. 2.0 (2016-08-03): https://cdn.clinicaltrials.gov/large-docs/41/NCT02199041/Prot_SAP_003.pdf